CLINICAL TRIAL: NCT01985126
Title: An Open-label, Multicenter, Phase 2 Trial Investigating the Efficacy and Safety of Daratumumab in Subjects With Multiple Myeloma Who Have Received at Least 3 Prior Lines of Therapy (Including a Proteasome Inhibitor and IMiD) or Are Double Refractory to a Proteasome Inhibitor and an IMiD
Brief Title: An Efficacy and Safety Study of Daratumumab in Patients With Multiple Myeloma Who Have Received at Least 3 Prior Lines of Therapy (Including a Proteasome Inhibitor [PI] and Immunomodulatory Drug [IMiD]) or Are Double Refractory to a PI and an IMiD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR102651; 54767414MMY2002 (Other: Janssen Research & Development, LLC); 2013-000752-18 (EudraCT Number)
Record Dates: First submitted 2013-07-22; First posted 2013-11-15 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Daratumumab; Proteasome inhibitor; Immunomodulatory drug; IMiD
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Methylprednisolone; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): During Stage 1 of Part 1, participants will be randomized to receive daratumumab treatment regimens in Group A and Group B. If in Stage 1, 1 or both of the treatment groups is considered to be ineffective and/or not well tolerated, then that treatment group will be terminated. Participants in Group B will be given the option to cross over to Group A if the investigator deems it in the best interest of the participants.
  Interventions: Drug: Daratumumab 16 mg/kg (Part 1); Drug: Daratumumab 8 mg/kg (Part 1); Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Diphenhydramine
- Part 2 (Experimental): Based on the Part 1 response rate, Group A or B daratumumab treatment will be selected as the treatment regimen for participants enrolled in Part 2.
  Interventions: Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Daratumumab (Part 2)

INTERVENTIONS:
Drug: Daratumumab 16 mg/kg (Part 1) — Daratumumab 16 mg/kg administered at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter by intravenous infusion
  Arms: Part 1
Drug: Daratumumab 8 mg/kg (Part 1) — Daratumumab 8 mg/kg every 4 weeks (Q4W) continuously by intravenous infusion
  Arms: Part 1
Drug: Methylprednisolone — Administered in prophylactic doses intravenously (or equivalent in accordance with local standards) prior to and after study drug administration. Intravenous administration is preferred, but oral steroids may be substituted
Drug: Acetaminophen — 650 to 1000 mg administered in prophylactic doses by mouth prior to study drug administration.
Drug: Diphenhydramine — 25 to 50 mg administered in prophylactic doses by mouth (or equivalent in accordance with local standards) prior to and after study drug administration.
Drug: Daratumumab (Part 2) — Based on the Part 1 response rate, Group A or B treatment will be selected as the treatment regimen for participants enrolled in Part 2.
  Arms: Part 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 daratumumab treatment regimens in participants with multiple myeloma who have received at least 3 prior lines of therapy (including a proteasome inhibitor [PI] and immunomodulatory drug [IMiD]) or are double refractory to a PI and an IMiD.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study of daratumumab for the treatment of participants with multiple myeloma who have received at least 3 prior lines of therapy including a PI and an IMiD or whose disease is double refractory to both a PI and an IMiD. Up to approximately 150 participants are to be enrolled. The study includes screening, treatment, and follow-up phases. Participants will receive daratumumab by intravenous infusion (28-day cycles) until disease progression, unacceptable toxicity, or other protocol-defined reasons. For all study drug administrations, participants will receive pre- and post-infusion medications for the prevention of infusion related reactions. Follow-up will continue until death, loss to follow up, consent withdrawal for study participation, or study end, whichever occurs first. The study will consist of 2 sequential parts (Part 1 and Part 2). The purpose of Part 1 is to select a dose and schedule for Part 2 of the study. Assessment of tumor response and disease progression will be conducted according to IMWG response criteria. Serial pharmacokinetic blood samples and a pharmacogenomic blood sample will be collected. Safety will be monitored throughout the study. At the end of the study, participants who are benefiting from treatment with daratumumab will have the option to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma according to protocol-defined criteria
* Evidence of disease progression on the most recent prior treatment regimen based on International Myeloma Working Group criteria
* Eastern Cooperative Oncology Group performance status score of 0, 1, or 2
* Laboratory values and electrocardiogram within protocol-defined parameters at screening

Exclusion Criteria:

* Received daratumumab or other anti-CD38 therapies previously
* Nonsecretory multiple myeloma
* Previously received an allogenic stem cell transplant or has received an autologous stem cell transplantation within 12 weeks
* Exhibiting clinical signs of meningeal involvement of multiple myeloma
* Known chronic obstructive pulmonary disease, persistent asthma, or a history of asthma within 5 years
* Seropositive for human immunodeficiency virus, hepatitis B or antibodies to hepatitis B surface and core antigens, or hepatitis C
* Has plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (23):
- United States (15):
  - Duarte, California
  - Los Angeles, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Detroit, Michigan
  - New Brunswick, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Madison, Wisconsin
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Montreal, Quebec
- Spain (3):
  - Barcelona
  - Salamanca
  - Valencia

REFERENCES:
- [Derived] Li X, Dosne AG, Perez Ruixo C, Perez Ruixo JJ. Pharmacodynamic-Mediated Drug Disposition (PDMDD) Model of Daratumumab Monotherapy in Patients with Multiple Myeloma. Clin Pharmacokinet. 2023 May;62(5):761-777. doi: 10.1007/s40262-023-01232-8. Epub 2023 Apr 6. PMID 37022569
- [Derived] Usmani SZ, Nahi H, Plesner T, Weiss BM, Bahlis NJ, Belch A, Voorhees PM, Laubach JP, van de Donk NWCJ, Ahmadi T, Uhlar CM, Wang J, Feng H, Qi M, Richardson PG, Lonial S. Daratumumab monotherapy in patients with heavily pretreated relapsed or refractory multiple myeloma: final results from the phase 2 GEN501 and SIRIUS trials. Lancet Haematol. 2020 Jun;7(6):e447-e455. doi: 10.1016/S2352-3026(20)30081-8. PMID 32470437
- [Derived] Adams HC 3rd, Stevenaert F, Krejcik J, Van der Borght K, Smets T, Bald J, Abraham Y, Ceulemans H, Chiu C, Vanhoof G, Usmani SZ, Plesner T, Lonial S, Nijhof I, Lokhorst HM, Mutis T, van de Donk NWCJ, Sasser AK, Casneuf T. High-Parameter Mass Cytometry Evaluation of Relapsed/Refractory Multiple Myeloma Patients Treated with Daratumumab Demonstrates Immune Modulation as a Novel Mechanism of Action. Cytometry A. 2019 Mar;95(3):279-289. doi: 10.1002/cyto.a.23693. Epub 2018 Dec 11. PMID 30536810
- [Derived] Usmani SZ, Khan I, Chiu C, Foureau D, Druhan LJ, Rigby K, Casneuf T, Sasser AK. Deep sustained response to daratumumab monotherapy associated with T-cell expansion in triple refractory myeloma. Exp Hematol Oncol. 2018 Feb 7;7:3. doi: 10.1186/s40164-018-0096-7. eCollection 2018. PMID 29445583
- [Derived] Nijhof IS, Casneuf T, van Velzen J, van Kessel B, Axel AE, Syed K, Groen RW, van Duin M, Sonneveld P, Minnema MC, Zweegman S, Chiu C, Bloem AC, Mutis T, Lokhorst HM, Sasser AK, van de Donk NW. CD38 expression and complement inhibitors affect response and resistance to daratumumab therapy in myeloma. Blood. 2016 Aug 18;128(7):959-70. doi: 10.1182/blood-2016-03-703439. Epub 2016 Jun 15. PMID 27307294
- [Derived] Lonial S, Weiss BM, Usmani SZ, Singhal S, Chari A, Bahlis NJ, Belch A, Krishnan A, Vescio RA, Mateos MV, Mazumder A, Orlowski RZ, Sutherland HJ, Blade J, Scott EC, Oriol A, Berdeja J, Gharibo M, Stevens DA, LeBlanc R, Sebag M, Callander N, Jakubowiak A, White D, de la Rubia J, Richardson PG, Lisby S, Feng H, Uhlar CM, Khan I, Ahmadi T, Voorhees PM. Daratumumab monotherapy in patients with treatment-refractory multiple myeloma (SIRIUS): an open-label, randomised, phase 2 trial. Lancet. 2016 Apr 9;387(10027):1551-1560. doi: 10.1016/S0140-6736(15)01120-4. Epub 2016 Jan 7. PMID 26778538

RESULTS

PARTICIPANT FLOW:
Groups:
- Daratumumab 8 mg/kg: Daratumumab 8 milligram per kilogram (mg/kg) every 4 weeks (Q4W) until disease progression or unacceptable toxicity.
- Daratumumab 16 mg/kg: Daratumumab 16 mg/kg weekly for 8 weeks; then every 2 weeks (Q2W) for 16 weeks; then Q4W until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Started | 18 | 106
Completed | 0 | 0
Not Completed | 18 | 106
Not completed — Death | 15 | 69
Not completed — Lost to Follow-up | 0 | 8
Not completed — Study Terminated By Sponsor | 1 | 22
Not completed — Withdrawal by Subject | 2 | 7

BASELINE CHARACTERISTICS:
Population: All treated Analysis Set included all participants who received at least 1 dose of daratumumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg | Total
Number analyzed (Participants) | 18 | 106 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 58 | 66
  >=65 years | 10 | 48 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.72) | 62.9 (10) | 63.1 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 54 | 60
  Male | 12 | 52 | 64
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 22 | 22
  Spain | 3 | 9 | 12
  United States | 15 | 75 | 90
Stage of Disease (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) system consists of stage I: beta2-microglobulin less than (<)3.5 milligram per liter (mg/l) and albumin greater than or equal to (>=) 3.5 gram (g)/100 ml; stage II: neither stage I nor stage III and stage III: beta2-microglobulin >= 5.5 mg/l.
  Participants
    I | 2 | 26 | 28
    II | 8 | 40 | 48
    III | 8 | 40 | 48
Number of Prior Lines of Therapy [Count of Participants; unit: Participants]
  <= 3 Lines | 6 | 19 | 25
  > 3 Lines | 12 | 87 | 99
Refractory to Proteasome Inhibitor (PI)/ Immunomodulatory Drug (IMiD) [Count of Participants; unit: Participants]
  Both a PI and IMiD | 15 | 101 | 116
  PI only | 1 | 3 | 4
  IMiD only | 0 | 1 | 1
  None | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response
Description: Overall response defined as percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). Per IMWG criteria, sCR: is defined as normal free light chain (FLC) ratio, and absence of clonal plasma cells (PCs) by immunohistochemistry, immunofluorescence or 2- to 4-color flow cytometry; CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5 % plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >= 90% reduction in serum M-protein plus urine M-protein level < 100mg/24 hours; PR: >= 50 % reduction of serum M-protein and reduction in 24 hour urinary M-protein by >= 90% or to <200 mg/24 hours; if the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria.
Time Frame: Up to 14.4 Months
Population: All treated analysis set included all participants who received at least 1 dose of daratumumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 18 | 106
percentage of participants | 11.1 [1.4 to 34.7] | 29.2 [20.8 to 38.9]

2. Secondary Outcome: Duration of Response
Description: Duration of response was calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in IMWG criteria. Disease progression (IMWG criteria): increase of 25 percent (%) from lowest response level in Serum M-component (the absolute increase must be >=0.5 g/dL) and/or; urine M-component (the absolute increase must be >=200 mg/24 hours) and/or; only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels (absolute increase must be >10 milligram per deciliter (mg/dL); Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.65 millimole per liter [mmol/L]) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: Up to 14.4 Months
Population: Responders in all treated analysis set. Only those participants with confirmed PR and those who experienced progressive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 2 | 31
months | NA [1.8 to NA] — These were Kaplan-Meier estimates. Median and/or upper limit of CI was not estimable because a small proportion of responders either progressed or died due to progressive disease. | 7.4 [5.5 to NA] — These were Kaplan-Meier estimates. Median and/or upper limit of CI was not estimable because a small proportion of responders either progressed or died due to progressive disease.

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the number of days from administration of the first infusion (Day 1) to date of death. Median Overall Survival was estimated by using the Kaplan-Meier method.
Time Frame: Approximately up to 3 years
Population: All treated analysis set included all participants who received at least 1 dose of daratumumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 18 | 106
months | 19.45 [7.72 to 26.81] | 18.60 [13.67 to 25.00]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit rate defined as percentage of participants who achieved minimal response (MR) or better. MR: >=25% but <= 49% reduction of serum M-protein and reduction in urine M-protein by 50%-89%. If present at baseline 25% to 49% reduction in size of soft tissue plasmacytomas.
Time Frame: Up to 14.4 Months
Population: All treated analysis set included all participants who received at least 1 dose of daratumumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 18 | 106
percentage of participants | 22.2 [6.4 to 47.6] | 34.0 [25.0 to 43.8]

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the date of first dose of daratumumab to the date of initial documentation of a response (PR or better).
Time Frame: Up to 14.4 Months
Population: Responders in all treated analysis set. Only those participants with confirmed PR were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 2 | 31
months | 0.99 [0.95 to 1.02] | 0.99 [0.9 to 5.6]

6. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was defined as the time between the date of first dose of daratumumab and either disease progression or death, whichever occurs first.
Time Frame: Up to 14.4 Months
Population: All treated analysis set included all participants who received at least 1 dose of daratumumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 18 | 106
months | 4.86 [1.84 to NA] — Upper limit of CI was not estimable due to the relatively short duration of follow-up. | 3.65 [2.76 to 4.63]

7. Secondary Outcome: Time to Disease Progression
Description: Time to progression was defined as the number of days from the date of first dose of daratumumab to the date of first record of disease progression.
Time Frame: Up to 14.4 Months
Population: All treated analysis set included all participants who received at least 1 dose of daratumumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 18 | 106
months | 4.86 [1.84 to NA] — Upper limit of CI was not estimable due to the relatively short duration of follow-up. | 3.71 [2.79 to 5.39]

ADVERSE EVENTS:
Time Frame: Approximately up to 3.8 years
Description: All treated Analysis Set included all participants who received at least 1 dose of daratumumab.
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Serious Adverse Events (participants affected / at risk) | 6/18 | 33/106
Other Adverse Events (participants affected / at risk) | 18/18 | 105/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab 8 mg/kg (N=18) | Daratumumab 16 mg/kg (N=106)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Faecal Incontinence (Gastrointestinal disorders) | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 5
Pyrexia (General disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
H1n1 Influenza (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 2
Parainfluenzae Virus Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4
Pneumonia Streptococcal (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Oxygen Saturation Abnormal (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Plasma Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab 8 mg/kg (N=18) | Daratumumab 16 mg/kg (N=106)
Anaemia (Blood and lymphatic system disorders) | 9 | 39
Leukopenia (Blood and lymphatic system disorders) | 2 | 8
Lymphopenia (Blood and lymphatic system disorders) | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 28
Sinus Tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 3
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0
Ear Discomfort (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 3
Abdominal Distension (Gastrointestinal disorders) | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 7
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 19
Diarrhoea (Gastrointestinal disorders) | 4 | 22
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 34
Vomiting (Gastrointestinal disorders) | 2 | 19
Asthenia (General disorders) | 2 | 12
Chest Discomfort (General disorders) | 1 | 3
Chills (General disorders) | 6 | 10
Fatigue (General disorders) | 6 | 42
Non-Cardiac Chest Pain (General disorders) | 1 | 6
Oedema (General disorders) | 1 | 2
Oedema Peripheral (General disorders) | 2 | 9
Pain (General disorders) | 1 | 6
Pyrexia (General disorders) | 5 | 20
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 7
Candida Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 4
Nasopharyngitis (Infections and infestations) | 1 | 8
Pneumonia (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 1 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 21
Urinary Tract Infection (Infections and infestations) | 0 | 7
Contusion (Injury, poisoning and procedural complications) | 1 | 5
Aspartate Aminotransferase Increased (Investigations) | 1 | 4
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 4
Blood Creatinine Increased (Investigations) | 7 | 9
Blood Urea Increased (Investigations) | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 1
Transaminases Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 2 | 5
Weight Increased (Investigations) | 1 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 19
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 20
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 25
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 10
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 9
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 15
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 20
Anaesthesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 10
Dysgeusia (Nervous system disorders) | 2 | 3
Encephalopathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 13
Hypoaesthesia (Nervous system disorders) | 1 | 6
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 6
Sciatica (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 0 | 8
Confusional State (Psychiatric disorders) | 1 | 7
Depression (Psychiatric disorders) | 1 | 3
Mental Status Changes (Psychiatric disorders) | 1 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 2
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 1
Nipple Pain (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 18
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 22
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 8 | 12
Hypotension (Vascular disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.